CLINICAL TRIAL: NCT05429775
Title: A Single Part, Four Period Sequential, Open Label Study Designed to Evaluate the In Vivo Performance of Oral Liquid Formulations of Budesonide in the Fasted State in Healthy Subjects
Brief Title: In Vivo Performance of Oral Liquid Formulations of Budesonide in the Fasted State in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SAN-0385/1828-BUD-3
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Budesonide: Formulation 1 (Experimental): single dose of 2 mg oral suspension formulation 1 administered orally under fasting conditions
  Interventions: Drug: Budesonide
- Budesonide: Formulation 2 (Experimental): single dose of 2 mg oral suspension formulation 2 administered orally under fasting conditions
  Interventions: Drug: Budesonide
- Budesonide: Formulation 3 (Experimental): single dose of 2 mg oral suspension formulation 3 administered orally under fasting conditions
  Interventions: Drug: Budesonide
- Budesonide: Formulation 4 (Experimental): single dose of 2 mg oral suspension formulation 4 administered orally under fasting conditions
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — single dose of 2 mg oral suspension formulation administered orally under fasting conditions

SUMMARY:
This is a single centre, open-label, sequential, single dose 4-period crossover, scintigraphic imaging study in healthy male and non-pregnant, non-lactating female subjects.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. For each treatment period, subjects will be admitted to the clinical unit on the evening prior to IMP administration (Day -1) and will fast overnight for a minimum of 8 h. On the morning of Day 1, subjects will receive IMP in the fasted state and will remain on site until 24 h post-dose. Following Period 2, there will be an interim analysis and review of safety and scintigraphy data from dosed regimens in order to determine which formulations will be used in subsequent periods. A follow-up phone call will take place 3 to 5 days post-final dose to ensure the ongoing wellbeing of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 30 to 65 years
* Body mass index 18.0 to 32.0 kg/m2

Exclusion Criteria:

* None

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Total oesophageal transit time | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.
Time at which 10% radiolabel administered has arrived in the oesophagus from the mouth (T10%) (min) | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.
Time at which 50% radiolabel administered has arrived in the oesophagus from the mouth (T50%) (min) | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.
Time at which the amount of radiolabel present in the oesophagus peaks (Tmax) (min) | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.
Time at which 90% of the radiolabel present at Tmax has left the oesophagus (T90%) (min) | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.
Total amount of radiolabel present in the oesophagus and the three regions over time | During procedure
  A comparison of the in vivo oesophageal transit times of budesonide suspension formulations will be determined using scintigraphic methods.

SECONDARY OUTCOMES:
Number of adverse events | throughout the study, approximately 13 weeks
  Number of adverse events will be provided to get additional information on the safety and tolerability of budesonide suspension formulations after oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (1):
- Sandoz Investigative Site, Nottingham, England, United Kingdom